CLINICAL TRIAL: NCT04166786
Title: Steroid Profile: Differentiating Testosterone Administration From (Simultaneous) Ethanol Consumption: Evaluation of Newly Developed Markers
Brief Title: Steroid Profile: Differentiating Testosterone Administration From (Simultaneous) Ethanol Consumption
Acronym: SPOL1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: IMIMFTCL/SPOL/1
Record Dates: First submitted 2019-11-07; First posted 2019-11-18 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-09

CONDITIONS: Healthy Volunteers
Keywords: Testosterone; Ethanol; Anti-doping control; Athletic performance
MeSH Terms: interventions — Petrolatum

STUDY DESIGN:
Intervention Model Description: Subjects receive 4 different treatment conditions (testosterone+ethanol placebo, ethanol+testosterone placebo, testosterone+ethanol, and placebo testosterone+placebo ethanol), separated by a wash-out period of 15 days. The order of the treatment conditions is randomly assigned.
Who Masked: Participant
Masking Description: Placebo treatments are administered in the same posology as active treatments (testosterone and ethanol).
  Ethanol is diluted in placebo (lemon-flavoured water) to prevent differentiation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Testosterone + Ethanol (Experimental): Subjects receive a 3-day treatment with testosterone in combination with ethanol consumption. Subjects have to collect urine in different fractions until 48h post-administration. Blood and saliva samples are also obtained.
  Interventions: Drug: Testosterone gel; Drug: Ethanol Solution
- Testosterone placebo + Ethanol (Other): Subjects receive a 3-day treatment with testosterone placebo (vaseline) in combination with ethanol consumption. Subjects have to collect urine in different fractions until 48h post-administration. Blood and saliva samples are also obtained.
  Interventions: Drug: Ethanol Solution; Drug: Testosterone placebo (vaseline)
- Testosterone + Ethanol placebo (Other): Subjects receive a 3-day treatment with testosterone in combination with ethanol placebo (lemon-flavoured water). Subjects have to collect urine in different fractions until 48h post-administration. Blood and saliva samples are also obtained.
  Interventions: Drug: Testosterone gel; Drug: Ethanol placebo (lemon-flavoured water)
- Testosterone placebo + Ethanol placebo (Placebo Comparator): Subjects receive a 3-day treatment with testosterone placebo (vaseline) in combination with ethanol placebo (lemon-flavoured water). Subjects have to collect urine in different fractions until 48h post-administration. Blood and saliva samples are also obtained.
  Interventions: Drug: Testosterone placebo (vaseline); Drug: Ethanol placebo (lemon-flavoured water)

INTERVENTIONS:
Drug: Testosterone gel — Subjects receive a daily transdermal dose of 100 mg of testosterone (2 sachets of 5 g of gel) during 3 days.
  Other Names: Testogel 50 mg®
  Arms: Testosterone + Ethanol; Testosterone + Ethanol placebo
Drug: Ethanol Solution — Subjects receive a daily administration of 30 g of ethanol (94 mL of Vodka Absolut® diluted in 300 mL of lemon-flavoured water Fontvella®) during 3 days.
  Other Names: Vodka Absolut®
  Arms: Testosterone + Ethanol; Testosterone placebo + Ethanol
Drug: Testosterone placebo (vaseline) — Subjects receive a daily transdermal dose of 5 g of pure vaseline ointment during 3 days.
  Other Names: Vaselina Pura Pege®
  Arms: Testosterone placebo + Ethanol; Testosterone placebo + Ethanol placebo
Drug: Ethanol placebo (lemon-flavoured water) — Subjects receive a daily administration of 394 mL of lemon-flavored-water Fontvella® during 3 days.
  Other Names: Lemon flavored-water Fontvella®
  Arms: Testosterone + Ethanol placebo; Testosterone placebo + Ethanol placebo

SUMMARY:
Background:

Testosterone is an anabolic steroid widely known to improve physical performance. Its consumption is banned by the World Anti-Doping Agency (WADA). The steroid profile is one of the components of the Athlete's Biological Passport (ABP), which consists of selected biological variables that indirectly reveal the effects of doping. Alcohol consumption has been proved to alter the steroid profile and this may lead to the use of ethanol as a masking agent for testosterone administration.

Hypothesis:

Ratios of different testosterone biomarkers vary after ethanol administration: [6-hydroxy-androsterone-3-glucuronide (6OH-Andros3G) / epitestosterone-glucuronide (EG)] and [6-hydroxy-etiocholanolone-3-glucuronide (6OH-Etio3G) / EG] decrease, while [testosterone-glucuronide (TG) / EG] increases.

Primary objective:

To evaluate if the combination of the markers TG, EG, 6OH-Andros3G and 6OH-Etio3G, as well as ethyl glucuronide (EtG) and ethyl sulfate (EtS), can be routinely used to differentiate between changes in the steroid profile due exclusively to the consumption of alcohol and those produced when alcohol is consumed during a testosterone administration.

Secondary objectives:

1. To explore the potential of the simultaneous determination of both phase I and phase II metabolites in alternative matrices (plasma from blood samples collected as for the haematological module of ABP, or saliva) in the screening of testosterone misuse.
2. To look for the differences into a comprehensive steroid profile (determined in urine, plasma and saliva) between samples collected after testosterone administration and after the combination of testosterone and ethanol.

Methods:

Phase I, single-blind, crossover-design clinical trial, placebo controlled, with 4 conditions randomly assigned in male healthy caucasian subjects with a wash-out period between treatments.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Caucasian men aged 18 to 40 years.
* Clinical history and physical examination demonstrating no organic or psychiatric disorders.
* The ECG and general blood and urine laboratory tests performed before the study should be within normal ranges. Minor or occasional changes from normal ranges are accepted if, in the investigator's opinion, considering the current state of the art, they are not clinically significant, are not life-threatening for the subjects and do not interfere with the product assessment. These changes and their non-relevance will be justified in writing specifically.
* The body mass index (BMI=weigh/height2) will range from 19 to 27 kg/m2, and the weight from 50 to 100 kg.
* Understanding and accepting the study procedures and signing the informed consent.
* Agreeing to follow a diet free from ethanol in the 72 hours prior to the start of each session and until the end of the study.
* Subjects with social or recreational alcohol consumption, at least 3 Standard Drink/week and subjects with experience in several drunkenness.
* Volunteers with normal steroidal profile for Caucasian population (0.7 ≤T / E ≤3)

Exclusion Criteria:

* Not meeting the inclusion criteria.
* Allergy, idiosyncrasy, hypersensitivity or adverse reactions to the active substance of Testogel gel®, which is synthesized from soy, or to any of the excipients or to vaseline ointment.
* Subjects with intolerance or adverse reactions to ethanol.
* History or clinical evidence of alcoholism, drug abuse, or regular use of psychoactive drugs.
* History or clinical evidence of cardiovascular, respiratory, renal, hepatic, endocrine, gastrointestinal, hematological, neurological, dermatological or other acute or chronic diseases that, in the opinion of the Principal Investigator or the collaborators designated by it, may pose a risk to the subjects or interfere with the objectives of the study. Especially history of epilepsy and migraine, edema, hypertension, diabetes mellitus, hypercalcemia or polyglobulia.
* History of psychiatric disorders.
* History or clinical evidence of gastrointestinal, liver, renal or other disorders which may lead to suspecting a disorder in drug absorption, distribution, metabolism or excretion, or that suggest gastrointestinal irritation due to drugs.
* Subjects with contraindications to treatment with the study drugs (according to the respective technical data sheets). Especially a history of breast cancer, liver cancer, suspicion or confirmation of prostate carcinoma Subjects and subjects who have suffered a hospitalization caused by alcohol intoxication or who have received treatment for drunkenness
* Having suffered any organic disease or major surgery in the three months prior to the study start.
* Symptoms compatible with a prostatic syndrome: increase in the number of urinations, difficulty to initiate urination, thinner and less potent urine stream, urination in several times, incomplete emptying of urine feeling.
* Prostate-specific antigen (PSA) values outside the normal range for the volunteer's age.
* Subjects with positive serology to Hepatitis B, C or HIV.
* Presence of bacterial, fungal or deep cuts in the area of skin chosen for cutaneous applications.
* Regular use of any drug in the month prior to the study sessions. The treatment with single or limited doses of symptomatic medicinal products in the week prior to the study sessions will not be a reason for exclusion if it is calculated that it has been cleared completely the day of the experimental session.
* Blood donation 8 weeks before or participation in other clinical trials with drugs in the previous 12 weeks.
* Smokers of more than 20 cigarettes per day.
* Taking more than 40 g of alcohol a day
* Consumers of more than 5 coffees, teas, cola drinks, or other stimulant drinks or with xanthines daily in the 3 months prior to the start of the study.
* Ingestion of vitamin supplements or antioxidants or Non-Steroidal Anti-Inflammatory Drugs (NSAID) in the two weeks preceding the study.
* Subjects unable to understand the nature, consequences of the study and the procedures requested to be followed.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2019-05-06 (Actual); Primary Completion 2019-09-26 (Actual); Study Completion 2019-09-26 (Actual)

PRIMARY OUTCOMES:
Change in steroid profile in urine | From baseline (pre-administration) to 48 hours after last administration (fractions: 0-2, 2-4, 4-6, 6-8, 8-24 hours each day, and 24-48 hours post-administration last day)
  Variation of the concentration of different endogenous steroids (testosterone, epitestosterone, androsterone, etiocholanolone, 3a,5a-androstanediol, 3a,5b-androstanediol, DHEAS, 5PTS, 5PDS, PTG, PDG) in urine before and after treatment administration.
Change in new steroid profile markers in plasma | From baseline (pre-administration) to 8 hours post-administration (at 0, 2, 4, 6, 8 hours each day)
  Variation of the concentration of new steroid profile markers (6OH-Andros3G, 6OH-Etio3G, testosterone free TG, Andros, Andros3G, Etio, Etio3G) in plasma before and after treatment administration.
Change in new steroid profile markers in saliva | From baseline (pre-administration) to 8 hours post-administration (at 0, 2, 4, 6, 8 hours each day)
  Variation of the concentration of new steroid profile markers (6OH-Andros3G, 6OH-Etio3G, testosterone free TG, Andros, Andros3G, Etio, Etio3G) in saliva before and after treatment administration.
Change in Ethyl glucuronide in urine | From baseline (pre-administration) to 48 hours post-administration (fractions: 0-2, 2-4, 4-6, 6-8, 8-24, 24-48 hours)
  Variation of the concentration of Ethyl glucuronide in urine before and after treatment administration.
Change in Ethyl sulfate in urine | From baseline (pre-administration) to 48 hours post-administration (fractions: 0-2, 2-4, 4-6, 6-8, 8-24, 24-48 hours)
  Variation of the concentration of Ethyl sulfate in urine before and after treatment administration.

CONTACTS AND LOCATIONS:
Overall Officials: Ana M Aldea Perona, Dr, Principal Investigator — IMIM (Hospital del Mar Medical Research Institute)
Locations (1):
- IMIM (Hospital del Mar Medical Research Institute), Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No